CLINICAL TRIAL: NCT05691075
Title: Metatarsophalangeal Arthrodesis of the Hallux : Observational Study Evaluating the Efficacy and Tolerance of Synthetic Methods Using Dorsal Plate and Large-diameter Screws
Brief Title: Metatarsophalangeal Arthrodesis of the Hallux
Acronym: ARTHRODESE
Status: Terminated | Type: Observational
Why Stopped: only 3 patients were included in this study
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A02518-35
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hallux Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metatarsophalangeal arthrodesis of the hallux with large diameter screws: Patient who can benefit from first-line arthrodesis using large-diameter screws
  Interventions: Procedure: Arthrodesis of the metatarsophalangeal joint
- Metatarsophalangeal arthrodesis of the hallux by plate: Patient who can benefit from a first intention arthrodesis by dorsal plate
  Interventions: Procedure: Arthrodesis of the metatarsophalangeal joint

INTERVENTIONS:
Procedure: Arthrodesis of the metatarsophalangeal joint — Isolated surgery of the first ray of hallux valgus, hallux varus or hallux rigidus by percutaneous or conventional approach

SUMMARY:
The purpose of the study is to describe the rate of bone fusion (radiological consolidation) in the 2 groups (A and B) 4 months after the operation.

DETAILED DESCRIPTION:
The main objective of the study is to describe the rate of bone fusion obtained with the different types of osteosynthesis material: dorsal plate, large-diameter compression screw.

Patients will be divided into two groups:

* patient undergoing arthrodesis of the hallux with a large diameter screw (group A)
* patient undergoing arthrodesis of the hallux by plate (group B)

This is a prospective, cross-sectional, open, comparative, non-randomized, non-interventional, monocentric study on two methods of synthesis (large-diameter plate or screw) of hallux metatarsophalangeal arthrodesis. Patients will be managed in accordance with current practice, the choice of surgical strategy (percutaneous / open) being left to the discretion of the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing isolated first ray surgery (M1 only) of hallux valgus, hallux varus or hallux rigidus by percutaneous or conventional approach;
* Patient who can benefit from first-line arthrodesis using a dorsal plate or large-diameter screw;
* Patient able to understand information related to the study and complete quality of life questionnaires;
* Patient accepting study follow-up visits;
* Patient having been informed and agreeing to participate in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Patient undergoing lateral ray surgery;
* Patient undergoing revision arthrodesis;
* Patient with a loss of bone substance requiring a graft;
* Patient suffering from chronic inflammatory disease;
* Patient treated with long-term immunosuppressive or corticosteroid treatments;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who can benefit from first-line arthrodesis using a dorsal plate or large-diameter screw.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Rate of bone fusion obtained with different types of osteosynthesis material (dorsal plate and large-diameter compressive screw) | 4 months
  Rate of bone fusion (radiological consolidation) in the 2 groups (A and B) 4 months after the operation, obtained with different types of osteosynthesis material: dorsal plate and large-diameter compressive screw

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Blomet, Paris, France

IPD SHARING:
Plan to Share IPD: No